CLINICAL TRIAL: NCT05138120
Title: Evaluating an Online Single-session Intervention (COMET) for Indian College Students
Brief Title: COMET India Follow-up Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 849593
Record Dates: First submitted 2021-11-16; First posted 2021-11-30 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2021-11

CONDITIONS: Depressive Symptoms; Anxiety; Happiness
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Common Elements Toolbox (Experimental)
  Interventions: Behavioral: Common Elements Toolbox
- Wait-list control (No Intervention)

INTERVENTIONS:
Behavioral: Common Elements Toolbox — An unguided online single-session intervention with four modules: behavioral activation, cognitive restructuring, gratitude, and self-compassion.
  Arms: Common Elements Toolbox

SUMMARY:
We are evaluating an online single-session intervention for mental health promotion among Indian college students.

ELIGIBILITY:
Inclusion Criteria:

* College Student
* Access to internet
* Proficient in English

Exclusion Criteria:

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-20 (Estimated); Primary Completion 2022-11-20 (Actual); Study Completion 2022-11-20 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ-9) | Up to 8 weeks post-intervention
  Depression questionnaire. Scores range from 0 to 27. Lower scores indicate less depression.
Change in Generalized Anxiety Disorder Screener-7 (GAD-7) | Up to 8 weeks post-intervention
  Anxiety questionnaire. Total scores range from 0-21. Lower scores indicate less anxiety.
Change in the Short Warwick-Edinburgh Mental Well-being Scale (SWEMWBS) | Up to 8 weeks post-intervention
  Well-being questionnaire. Total scores range from 7 to 35. Higher values indicate higher well-being scores.

SECONDARY OUTCOMES:
Ratings on the Acceptability of Intervention Measure (AIM) | Immediately after the intervention
  Questionnaire measuring the acceptability of an intervention. Acceptability refers to the perception that a given treatment is agreeable or satisfactory. The total score ranges from 4 to 20. Higher scores indicate higher acceptability ratings.
Ratings on the Intervention Appropriateness Measure (IAM) | Immediately after the intervention
  Questionnaire measuring the appropriateness of an intervention. Appropriateness refers to the perceived fit or relevance of an intervention. The total score ranges from 4 to 20. Higher scores indicate higher appropriateness.
Mechanisms of Change | Up to 8 weeks post-intervention
  Participants answered questions relating to each module's mechanism of change on a 7-point Likert Scale, from "strongly disagree" to "strongly agree".
  Specifically, we asked participants:
  How capable they feel about managing negative thoughts; If they will intentionally spend time doing activities they enjoy; If they will notice and appreciate good things; If they will
Secondary Control | Up to 8 weeks post-intervention
  We asked participants three items to assess secondary control (Weisz et al., 2010). The items are scored on a 4-point Likert scale, ranging from 0 ("Very false") to 3 ("Very true").
  The three items are:
  When something bad happens, I can find a way to think about it that makes me feel better.
  After a really hard day, I can make myself feel better by remembering some good things that happened.
  When bad things happen to me that I can't control, there are lots of things I can do to feel better.
  Higher scores indicate greater secondary control.
Positive and Negative Affect Schedule | Up to 8 weeks post-intervention
  Questionnaire measuring positive affect and negative affect. Scores on the positive affect subscale range from 10-50, with higher scores representing higher levels of positive affect. Scores on the negative affect subscale range from 10-50, with lower scores representing lower levels of negative affect.
Perceived Stress Scale-4 | Up to 8 weeks post-intervention
  Questionnaire measuring perceived stress. Scores range from 0-16, with higher scores indicating greater stress.